CLINICAL TRIAL: NCT04543214
Title: Outcome of Enhanced Recovery After Surgery (ERAS) Protocols in Patients Undergoing Small Bowel Surgery
Status: Completed | Type: Observational
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Principal Investigator, Services Hospital, Lahore
Other Study IDs: s15
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Enhanced Recovery After Surgery
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Enhanced recovery after surgery — Enhanced recovery after surgery (ERAS) protocols are multimodal perioperative care pathways designed to achieve early recovery after surgical procedures by maintaining preoperative organ function and reducing the profound stress response after surgery. It benefits patient by reducing complications and enhancing recovery and saves resources for the health care system. In this concept, surgeons work collaboratively with anesthesiologist, nurses, nutritionists and physical therapists to develop and manage the perioperative care.

SUMMARY:
It was a descriptive case series conducted it Department of Surgery, Services Hospital, Lahore. Total of 140 patients who underwent small bowel resection anastomosis were subjected to ERAS protocols.The objective of this study was to determine the outcome of applying enhanced recovery after surgery (ERAS) protocols in patients undergoing small bowel surgery.

DETAILED DESCRIPTION:
It was a descriptive case series study conducted at Surgical Unit II, Services Hospital, Lahore. Sample size of 140 cases was calculated with 95% confidence level, 4.5% margin of error while taking expected percentage of anastomotic leakage in 8% cases passed through Enhanced Recovery after Surgery protocole.9 Patients were selected by Non-probability Purposive Sampling. Patients of both sex groups with ages between 20-45 years. Having elective surgery of small bowel resection and anastomosis admitted through OPD were included in the study. Patient with co-morbid conditions falling in ASA Class III or greater and patients with metastatic tumours of small bowel were excluded from the study. 140 patients presenting in the surgical outdoor of Services Hospital, Lahore who fulfilled the inclusion criteria were included in the study. A detailed history was taken including demographic data (age, gender and address). Patients were requested to sign an informed consent after explaining them the details of the study. ERAS protocols were implemented. Patients were followed after 4 weeks post-operatively in outdoor and outcome were measured in terms of length of hospital stay, post-operative wound infection, anastomotic leakage and death. All the surgeries and the follow ups were performed by the consultant in charge of the unit to eliminate bias. Confounding variables were controlled by exclusion. All the data was recorded into the attached proforma.(annexed). All the collected data was entered into SPSS version 10. Numerical variables like age and length of hospital stay have been presented by mean ±SD. Categorical variables i-e gender, post-operative wound infection, anastomotic leakage and mortality have been presented by frequency and percentage. Data has been stratified for anastomotic leakage to deal with effect modifier. Chi square test has been applied post stratification with P-value ≤0.05 taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery of small bowel resection
* Benign and malignant non metastatic disease
* ASA-I and ASA-II patients

Exclusion Criteria:

* Uncontrolled diabetes
* Metastatic disease
* Malnourished patients
* Chronic renal Failure
* Chronic liver disease

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sample size of 140 cases was calculated with 95% confidence level, 4.5% margin of error while taking expected percentage of anastomotic leakage in 8% cases passed through Enhanced Recovery after Surgery protocole.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | 2 weeks
  Number of days patients stays in hospital
Postoperative wound infection | 2 weeks
  Number of patients developing erythema and purulent discharge from wound site
Anastomotic leakage | 4 weeks
  Number of patients developing leak from anastomotic site

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No